CLINICAL TRIAL: NCT06092684
Title: A Multicenter, Randomized, Double-blind Clinical Trial to Evaluate the Efficacy and Safety of BT-KTM-I Versus Ketanest® S for General Anesthesia in Elective Laparoscopic Surgery
Brief Title: The Efficacy and Safety of Esketamine in Elective Laparoscopic Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chengdu Brilliant Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BT-KTM-I-III-01
Record Dates: First submitted 2023-09-21; First posted 2023-10-23 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Laparoscopy; Anesthesia, Intravenous
MeSH Terms: interventions — Esketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BT-KTM-I (Experimental): Patients received 0.5mg/kg BT-KTM-I during anesthesia induction period. Patients received 0.5mg/kg/h BT-KTM-I during anesthesia maintenance period.
  Interventions: Drug: BT-KTM-I
- Ketanest®S (Active Comparator): Patients received 0.5mg/kg Ketanest®S during anesthesia induction period. Patients received 0.5mg/kg/h Ketanest®S during anesthesia maintenance period.
  Interventions: Drug: Ketanest®S

INTERVENTIONS:
Drug: BT-KTM-I — The dosage for anesthesia induction period was 0.5mg/kg, and the dosage for anesthesia maintenance period was 0.5mg/kg/h.
  Other Names: Esketamine
  Arms: BT-KTM-I
Drug: Ketanest®S — The dosage for anesthesia induction period was 0.5mg/kg, and the dosage for anesthesia maintenance period was 0.5mg/kg/h.
  Other Names: Esketamine
  Arms: Ketanest®S

SUMMARY:
The objective is to evaluate the efficacy and safety of BT-KTM-I(Esketamine Hydrochloride Injection produced by Chengdu Brilliant Pharmaceutical Co., Ltd.) for general anesthesia, using the Originator drug Ketanest®S(Esketamine Hydrochloride Injection) as a positive control.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, positive drug parallel controlled clinical trial, planned to include 358 subjects, including 179 in the experimental group and 179 in the control group. The entire study was divided into a screening period, surgery day, and follow-up observation period. The dosage for anesthesia induction period was 0.5mg/kg, and the dosage for anesthesia maintenance period was 0.5mg/kg/h. The experiment used vital signs, physical examination, laboratory examination, 12-lead electrocardiogram examination, and adverse events/serious adverse events for safety evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Age range from 18 to 60 years old (including threshold), regardless of gender;
2. Patients undergoing elective general anesthesia laparoscopic surgery (only tracheal intubation mechanical ventilation), 1 hour ≤ expected anesthesia time ≤ 2.5 hours;
3. The American Society of Anesthesiologists (ASA) score of Class I or II;
4. 18kg/m2<BMI<30kg/m2;
5. The subjects understand the purpose and procedure of this experiment, voluntarily participate in this experiment, and sign a written informed consent form.

Exclusion Criteria:

1. Patients with contraindications to general anesthesia, or those who have had previous anesthesia accidents;
2. Known intolerance or allergy to ketamine hydrochloride, esketamine hydrochloride, propofol, rocuronium bromide, opioids, neostigmine, atropine, belladonnae alkaloids;
3. Long-term (continuous or intermittent) use of benzodiazepines sleeping pills, opioid analgesics, or use of narcotic analgesics within 24 hours before randomization or use of narcotic drugs within 7 days;
4. Have a history of increased intraocular pressure (such as glaucoma) or puncture eye injury;
5. Patients with a history of asthma;
6. Patients with mental system diseases (schizophrenia, mania, insanity, etc.) or cognitive disorders;
7. Patients with a history of craniocerebral injury, possible presence of intracranial hypertension, cerebral aneurysm, cerebrovascular accident, and central nervous system disease;
8. Have a serious history of cardiovascular diseases (such as myocardial ischemia, heart failure and severe arrhythmia); Angina pectoris (unstable angina) caused by insufficient blood supply to the coronary arteries of the heart, or myocardial infarction occurring within the first 6 months before screening;
9. Hypertensive patients with systolic blood pressure still ≥ 140mmHg and/or diastolic blood pressure still ≥ 90mmHg after treatment with antihypertensive drugs;
10. Diabetic patients whose blood glucose was not satisfactorily controlled (fasting blood glucose ≥11.1mmol/L during the screening period);
11. Severe lipid metabolism abnormalities (such as triglycerides>5mmol/L, diabetic hyperlipidemia, familial hypercholesterolemia, lipoid nephropathy, acute pancreatitis with hyperlipidemia, etc.);
12. Have a history of hyperthyroidism;
13. Have a history of drug use within 2 years before screening;
14. Individuals with a history of alcohol abuse within 2 years before screening. alcoholism is defined as drinking more than 14 units of alcohol per week (1 unit =360mL beer or 45mL spirits with 40% alcohol or 150mL wine) or acute alcoholism or alcohol dependence;
15. Participants in any clinical trial (defined as receiving the experimental drug or placebo) within 3 months prior to screening;
16. Patients with respiratory management difficulties as determined by the investigators (modified Markov score level Ⅳ);
17. Abnormal coagulation function (PT or PT-INR ≥ 1.5×ULN, APTT ≥ 1.5×ULN), or with bleeding tendency (such as active digestive ulcer) or undergoing thrombolytic or anticoagulant treatment;
18. Anemia or thrombocytopenia (PLT≤80×109/L, HGB≤90g/L);
19. Abnormal liver function [ALT and (or) AST≥1.5×ULN, TBIL≥1.5×ULN];
20. Abnormal renal function (BUN≥1.5×ULN; Cr≥1.2×ULN)
21. Pregnant or lactating women; Women or men with fertility are unwilling to use contraception between the screening period and the end of the trial;
22. Subjects who are deemed by the investigators to have any other unfavorable factors for participating in this clinical trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 358 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2024-03-19 (Actual); Study Completion 2024-03-19 (Actual)

PRIMARY OUTCOMES:
The awakening time from anesthesia | The time from discontinuing the use of anesthetics (propofol) to subjects waking up immediately after surgery (following instructions to open their eyes)

SECONDARY OUTCOMES:
Incidence of adverse reactions in the mental system | Within 60 minutes after the subject wakes up

CONTACTS AND LOCATIONS:
Overall Officials: Wen Ouyang, MD, Principal Investigator — The Third Xiangya Hospital of Central South University
Locations (12):
- China (12):
  - The First Affiliated Hospital of Jinan University, Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Guizhou Provincial People's Hospital, Guiyang, Guizhou
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Hunan Provincial Maternal and Child Health Care Hospital, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - The Second Hospital University of South China, Hengyang, Hunan
  - Pidu District People's Hospital, Chengdu, Chengdu, Sichuan
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - West China Second University Hospital, Sichuan University, Chengdu, Sichuan
  - The Second People's hospital of Neijiang, Neijiang, Sichuan
  - The Second People's Hospital of Yibin, Yibin, Sichuan